CLINICAL TRIAL: NCT07038473
Title: Islet Autoantibody Early Detection in At-risk Children/Adolescents to Predict Type 1 Diabetes: a Cohort Study in Gulf Countries
Brief Title: Early Detection of Type 1 Diabetes in First Degree Relatives of Type 1 Diabetes Patients (DETECT T1D GULF)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PIR18651; U1111-1319-5409 (Registry Identifier: ICTRP)
Record Dates: First submitted 2025-06-06; First posted 2025-06-26 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Children, adolescents and first-degree relatives of T1D probands (Other): Blood samples will be collected from the participants and autoantibody testing will be performed. For participants who test positive for any autoantibodies, another autoantibody test and HbA1C test and Oral Glucose Tolerance Test (OGTT) or CGM (Continuous Glucose Monitoring) will be performed
  Interventions: Procedure: Investigational Procedure

INTERVENTIONS:
Procedure: Investigational Procedure — It consists of prospective blood sample collection from children, adolescents and first-degree relatives of T1D probands.
  Study without any Investigational Medicinal Product (IMP) administration.

SUMMARY:
The aim of this research is to identify pre-symptomatic Type 1 Diabetes (T1D) in young children and adolescents who have first degree relatives with T1D. This protocol has been developed to address the growing need for standardized T1D screening, monitoring, and data collection in alignment with international recommendations. The study's estimated duration is 13 months and will consist of two visits: Visit 1 (screening visit) and Visit 2 (confirmatory visit).

ELIGIBILITY:
Inclusion Criteria:

* Children and adolescents, age 1.5 years to 18 years
* First degree relatives of T1D probands
* Parent or legal guardian signing an informed consent

Exclusion Criteria:

* Already developed clinical overt T1D
* Known diabetes of any kind (type 1, type 2, Maturity Onset Diabetes of the Young - MODY)
* Have a previous history of being treated with insulin

Ages: 18 Months to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 3500 (Estimated)
Dates: Start 2025-12-25 (Estimated); Primary Completion 2026-12-25 (Estimated); Study Completion 2026-12-25 (Estimated)

PRIMARY OUTCOMES:
Proportion of at-risk (first-degree) relatives of T1D probands who meet the diagnostic criteria for Stage 1 or Stage 2 T1D | At Baseline (screening visit) and in 3 months, at Visit 2 (confirmatory visit)
  Stage 1 is defined by the presence of two or more diabetes-related autoantibodies with normoglycemia.
  Stage 2 is characterized by the presence of two or more diabetes-related autoantibodies with dysglycemia (impaired fasting glucose or impaired glucose tolerance) but without clinical symptoms of diabetes

SECONDARY OUTCOMES:
Proportion of participants who meet the criteria for Stage 3 Type 1 Diabetes (T1D) diagnosis | At Baseline (screening visit) and in 3 months, at Visit 2 (confirmatory visit)
  Stage 3 is defined by the presence of two or more diabetes-related autoantibodies, abnormal blood glucose levels, and clinical symptoms of T1D, such as polyuria, polydipsia, weight loss, and fatigue
Refusal rate - ratio of patients proposed for screening who did not accept autoantibody testing and follow-up monitoring | At Baseline (screening visit)
Acceptance rate - ratio of patients proposed for screening who accepted autoantibody testing and follow-up monitoring | At Baseline (screening visit) and in 3 months, at Visit 2 (confirmatory visit)

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org